CLINICAL TRIAL: NCT02587390
Title: A Study to Evaluate the Effects of Gemcabene on the Steady-State Pharmacokinetics and Pharmacodynamics of Simvastatin in Healthy Volunteers
Brief Title: Effect of Gemcabene on the Pharmacokinetics of Simvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1027-008
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia
Keywords: Pharmacokinetics; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg
  Interventions: Drug: Gemcabene 900 mg; Drug: Simvastatin 80 mg
- Simvastatin 80 mg (Active Comparator): Simvastatin 80 mg
  Interventions: Drug: Simvastatin 80 mg

INTERVENTIONS:
Drug: Gemcabene 900 mg — 3x300 mg Gemcabene tablets orally once daily (QD) for 15 days
  Arms: Gemcabene 900 mg
Drug: Simvastatin 80 mg — 2x40 mg Simvastatin tablets orally once daily (QD) for 15 days

SUMMARY:
The purpose of this study is to determine the effect of gemcabene on the pharmacokinetics of simvastatin 80 mg.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* >18 years of age
* Body weight 45 kg or greater

Exclusion Criteria:

* If female, of childbearing potential or lactation
* History of significant adverse reaction to any fibrate lipid-lowering agent or HMG-CoA reductase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-05; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 15 days
  Cmax
Pharmacokinetics | 15 days
  Area Under the Curve (AUC)

SECONDARY OUTCOMES:
Adverse Events | 57 days
Clinical Laboratory - hematology, chemistry, urinalysis | 57 days
  Clinical Laboratory Abnormalities
ECG | 57 days
  Clinically Significant Changes